CLINICAL TRIAL: NCT02452723
Title: A Single Arm, Open-Label Phase 1 Study to Evaluate the Safety and Tolerability of ISC-hpNSC Injected Into the Striatum and Substantia Nigra of Patients With Parkinson's Disease
Brief Title: A Study to Evaluate the Safety of Neural Stem Cells in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyto Therapeutics Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISC-hpNSC
Record Dates: First submitted 2015-05-18; First posted 2015-05-25 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ISC-hpNSC (Experimental)
  Interventions: Biological: ISC-hpNSC

INTERVENTIONS:
Biological: ISC-hpNSC

SUMMARY:
This study will evaluate the safety of an investigational cell transplantation therapy, ISC-hpNSC, in patients with Parkinson's disease. All patients will receive the therapy, which consists of human neural stem cells. Three dose levels will be examined in the study.

DETAILED DESCRIPTION:
ISC-hpNSC is a cellular therapeutic consisting of human parthenogenetic neural stem cells (hpNSC). ISC-hpNSC will be injected intracerebrally to the striatum and substantia nigra of patients with Parkinson's disease (PD).

The study will enroll 4 patients for cell injection at each of three different doses. A total of 12 patients with moderate to severe PD will be treated. Each patient receives a single dose. The main objective of the study is to evaluate the safety of the cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF) indicating the patient has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts
* Patient diagnosed with idiopathic PD of ≤ 13 years duration, as defined by the United Kingdom (UK) Parkinson's Disease Society Brain Bank criteria
* Outpatients (male and female) 30 - 70 years old. Females must be of non-child bearing potential, or with a negative pregnancy test and not breast-feeding
* Patients receiving a stable dose of levodopa for at least 3 months with the expectation that the treatment will remain unchanged throughout the course of the patient's participation in the trial
* Patients receiving an anti-parkinsonian treatment at a stable dose for at least 3 months with the expectation that the treatment will remain unchanged throughout the course of the patient's participation in the trial
* Hoehn and Yahr stage II-IV during "ON" time
* Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) in the "OFF" state ≤ 49
* Positive dopaminergic response of ≥ 33% decrease in UPDRS motor scores between "OFF" and "ON" states at screening, and unequivocal clinical off periods
* Patient is experiencing motor fluctuations with at least two cumulative hours of daily "OFF" -time during the waking period, which is measured on at least two consecutive days
* History of anti-parkinsonian treatment with sufficient doses of levodopa
* Stable, well-controlled concomitant disorders that would not contraindicate general anesthesia or stereotactic neurosurgery
* No abnormalities on baseline brain MRI
* Insufficient control of PD symptoms or intolerable side effects with optimized oral PD therapy
* Montreal Cognitive Assessment (MOCA) score ≥ 26
* Willing to fully comply with all study procedures and requirements of the trial
* No surgery for PD or been treated with neuroleptics in the past 6 months except low-dose quetiapine fumarate or clozapine
* No significant further improvement with physical therapy/rehabilitation

Exclusion Criteria:

* Mild cognitive impairment of dementia (MOCA score < 26)
* The extent or severity of the disease is not measurable
* Severe dyskinesia in the "OFF" or "ON" states (violent dyskinesias, incompatible with any normal motor task)
* Pre-existing medical conditions such as bleeding disorders, septicemia, major cardiovascular, cerebrovascular or psychiatric disease
* Any current or relevant previous history of serious, severe or unstable physical or psychiatric illness or medical disorder that may make the participant unlikely to fully complete the study (depression, anxiety, cognitive impairment or impulse control disorder)
* Clinically significant abnormal hematologic evaluation (blood count, partial thromboplastin time (PTT)), blood chemistry (glucose, blood urea nitrogen (BUN), creatinine, electrolytes), liver function tests (aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGTP), total protein, bilirubin)
* Any active infectious disease of any nature, including clinically active viral infections (seropositive for Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV), Hepatitis B Virus (HBV) and Syphilis
* Severe obesity
* Previous intracranial surgery, including deep-brain stimulation
* History of seizures
* Substance abuse (recent history of alcohol abuse or other drugs such as barbiturates, cannabinoids and amphetamines)
* Use of anti-platelet agents or other anti-coagulants
* Signs of any malignant disease
* Any use of immunosuppressive drugs
* Enrollment in other investigational drug trial or has completed any trial within the last 3 months
* Patients that cannot undergo MRI or PET scanning (i.e. patients with implanted pacemakers)
* Patients unable to travel to the PET scanning center
* Any other condition which clinician regards as making patient unsuitable for trial

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2025-06-18 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs), serious TEAEs, related TEAEs, severe TEAEs | 12 month

SECONDARY OUTCOMES:
Change in UPDRS score from baseline | Baseline and 12 months
Proportion of patients with improvement defined as any reduction in UPDRS motor score | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Neurology, The Royal Melbourne Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Garitaonandia I, Gonzalez R, Sherman G, Semechkin A, Evans A, Kern R. Novel Approach to Stem Cell Therapy in Parkinson's Disease. Stem Cells Dev. 2018 Jul 15;27(14):951-957. doi: 10.1089/scd.2018.0001. PMID 29882481
- [Derived] Garitaonandia I, Gonzalez R, Christiansen-Weber T, Abramihina T, Poustovoitov M, Noskov A, Sherman G, Semechkin A, Snyder E, Kern R. Neural Stem Cell Tumorigenicity and Biodistribution Assessment for Phase I Clinical Trial in Parkinson's Disease. Sci Rep. 2016 Sep 30;6:34478. doi: 10.1038/srep34478. PMID 27686862
- [Derived] Gonzalez R, Garitaonandia I, Poustovoitov M, Abramihina T, McEntire C, Culp B, Attwood J, Noskov A, Christiansen-Weber T, Khater M, Mora-Castilla S, To C, Crain A, Sherman G, Semechkin A, Laurent LC, Elsworth JD, Sladek J, Snyder EY, Redmond DE Jr, Kern RA. Neural Stem Cells Derived from Human Parthenogenetic Stem Cells Engraft and Promote Recovery in a Nonhuman Primate Model of Parkinson's Disease. Cell Transplant. 2016 Nov;25(11):1945-1966. doi: 10.3727/096368916X691682. PMID 27213850